CLINICAL TRIAL: NCT01505270
Title: The Prevalence of Psychological and Medical Comorbidities Among Children Suffering From Autistic Spectrum Disorder and the Differences Between Ethnic Groups in Israel
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0103-11-HYMC
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Autistic Children
  Interventions: Other: Retrospective case study

INTERVENTIONS:
Other: Retrospective case study — Retrospective case study

SUMMARY:
It is known that several psychological and medical comorbidities are frequently found among children suffering from autistic spectrum disorders. Our aim is to investigate which comorbidities are most common among those children and whether there are differences among the different ethnic groups found in Israel.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with autism

Exclusion Criteria:

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of autistic children with comorbidities | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel